CLINICAL TRIAL: NCT03480932
Title: Role of Pegylated Interferon in Combination With Direct Acting Antivirals (DAAs) to Cure Hepatitis C As Soon As Possible (ASAP) - Hepatitis C [ASAP-C]
Brief Title: Role of Pegylated Interferon in Combination With DAAs to Cure Hepatitis C As Soon As Possible - Hepatitis C [ASAP-C]
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); YR Gaitonde Centre for AIDS Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA026727 (NIH); R01DA026727 (NIH)
Record Dates: First submitted 2018-01-29; First posted 2018-03-29 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C, Chronic
Keywords: directly observed therapy; sofosbuvir; daclatasvir; pegylated interferon; resource-limited setting
MeSH Terms: conditions — Hepatitis C, Chronic; Directly Observed Therapy | interventions — Sofosbuvir; daclatasvir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SOF+DAC+PEG (Active Comparator): Sofosbuvir (400mg/daily) + Daclatasvir (60mg/daily) + Pegylated Interferon alfa-2a (180µg/weekly) for 4 weeks with a field-based DOT approach
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir; Drug: Pegylated Interferon alfa-2a
- SOF+DAC, DOT (Active Comparator): Sofosbuvir (400mg/daily) + Daclatasvir (60mg/daily) for 12 weeks with a field-based DOT approach
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir
- SOF+DAC, standard (Active Comparator): Sofosbuvir (400mg/daily) + Daclatasvir (60mg/daily) for 12 weeks with standard of care dispensation (4 monthly doses)
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir

INTERVENTIONS:
Drug: Sofosbuvir — Direct acting antiviral agent used for the treatment of hepatitis C
  Other Names: Sovaldi; Hepcvir; MyHep; Hepcinat; Resof; SoviHep
Drug: Daclatasvir — Direct acting antiviral agent used for the treatment of hepatitis C
  Other Names: Daklinza; Natdac; Daclahep; Dacihep; Hepdac; Mydekla
Drug: Pegylated Interferon alfa-2a — Antiviral agent used for the treatment of hepatitis C
  Other Names: Pegasys; Taspiance
  Arms: SOF+DAC+PEG

SUMMARY:
The primary objective of this pilot trial is to compare the efficacy, measured as sustained virologic response (SVR) at least 12 weeks after completion of therapy, across three study regimens/delivery modalities: Arm 1 - 4 weeks of sofosbuvir (SOF) + daclatasvir (DAC) + pegylated interferon alfa-2a (PEG) delivered using directly observed therapy (DOT); Arm 2 - 12 weeks of SOF+DAC delivered using DOT; and Arm 3 - 12 weeks of SOF+DAC delivered as per standard of care (monthly dispensation with no DOT). Secondary objectives are 1)To compare the cost per SVR for each of the three study arms; 2) To compare adherence among persons across the three study arms; 3) To evaluate the safety, tolerability and acceptability of treatment in the three arms.

DETAILED DESCRIPTION:
This will be a non-blinded randomized clinical trial with 150 participants randomized at a 1:1:1 allocation ratio to one of three treatment arms.

Arm 1: Sofosbuvir (400mg/daily) + Daclatasvir (60mg/daily) + Pegylated Interferon alfa-2a (180µg/weekly) for 4 weeks with a field-based DOT approach

Arm 2: Sofosbuvir (400mg/daily) + Daclatasvir (60mg/daily) for 12 weeks with a field-based DOT approach

Arm 3: Sofosbuvir (400mg/daily) + Daclatasvir (60mg/daily) for 12 weeks with standard of care dispensation (4 monthly doses)

Pegylated-interferon alfa-2a (PEG) will be delivered subcutaneously once weekly. Sofosbuvir (SOF) and Daclatasvir (DAC) will be taken orally once daily for the entire study period.

The study will take place at the YR Gaitonde Centre for AIDS Education (YRG) and Johns Hopkins University (JHU) Collaborative Integrated Care Center (YRG-JHU ICC) located within the premises of the Chattisgarh Institute of Medical Sciences (CIMS) in Bilaspur in the state of Chattisgarh, India.

Participants will be recruited from the YRG-JHU ICC in Bilaspur, which currently has 514 registered HCV antibody positive clients. The Bilaspur ICC is in the Chattisgarh Institute for Medical Sciences (CIMS).

The primary outcome will be sustained virologic response (SVR12). Secondary outcomes include cost per SVR12, adherence, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Age ≥ 18 years
3. Documented evidence of chronic HCV infection (HCV RNA positive)
4. Participant is a resident of Bilaspur and can provide locator information that can be verified by one of the study staff
5. If participant is co-infected with HIV, he/she must have a cluster of differentiation 4 (CD4) > 350 cells/mm3 and be either: 1) antiretroviral therapy (ART) naïve or 2) on ART be on a tenofovir-containing regimen. If a subject's CD4 drops below 350 cells/μl (current threshold for HIV treatment in India), he/she will be able to initiate ART but we will ensure that the subject starts on a tenofovir-containing regimen, which is currently the standard for persons newly initiating ART in India.
6. Subjects must have the following laboratory parameters at screening:

   1. alanine aminotransferase (ALT) ≤ 10 x the upper limit of normal (ULN)
   2. aspartate aminotransferase (AST) ≤ 10 x ULN
   3. Hemoglobin ≥ 10 g/dl for male and 9 g/dl for female subjects
   4. International normalized ratio (INR) ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   5. Albumin ≥ 3 g/dl
   6. Direct bilirubin ≤ 1.5 x ULN
   7. Creatinine clearance ≥ 30 ml/min as calculated by the Cockcroft-Gault Equation
   8. Alpha fetoprotein < 50 ng/ml
   9. Absolute neutrophil count (ANC) ≥ 1,500/μL
   10. Platelets ≥ 90,000/μL
   11. Thyroid stimulating hormone (TSH) ≤ ULN
   12. FIB-4 <3.25. FIB-4 is a non-invasive Marker of Hepatic Fibrosis: Fibrosis-4 (FIB-4) which is calculated as the ratio of age in years and aminotransferase to platelet count. It is a non-invasive hepatic fibrosis index score combining standard biochemical values, platelets, alanine aminotransferase (ALT), AST and age that is calculated using formula: FIB-4 = (Age [years] x AST [U/L]) / (platelets [10^9/L] x (square root of ALT [U/L])). A FIB-4 index of < 1.45 indicated no or moderate fibrosis and an index of > 3.25 indicated extensive fibrosis/cirrhosis.) Participants with a FIB-4 >3.25 will be referred to the medical gastroenterology department for further assessment for cirrhosis. If cirrhosis is ruled out by medical gastroenterology, participants can be rescreened for the study.
7. A female subject is eligible to enroll in the study if it is confirmed that she is:

   1. Not pregnant or nursing
   2. Not of childbearing potential (i.e., women who have had a hysterectomy, have both ovaries removed or medically documented ovarian failure, or are postmenopausal women > 50 years of age with cessation (for ≥12 months) of previously occurring menses)
   3. Of childbearing potential (i.e., women who have not had a hysterectomy, both ovaries removed or medically documented ovarian failure). [NOTE: Women ≤50 years of age with amenorrhea will be considered to be of childbearing potential.] These women must have a negative urine pregnancy test at screening and a negative urine pregnancy test on the Baseline /Day 1 visit prior to randomization and agree to one of the following modes of contraception for the duration of treatment and 12 weeks thereafter.

      * Complete abstinence from intercourse. Periodic abstinence (e.g., calendar, ovulation, sumptothermal, post-ovulation methods) is NOT permitted.

   or

   i. Consistent and correct use of 1 of the following methods of birth control listed below in addition to a male partner who correctly uses a condom from 3 weeks prior to Baseline/Day 1 until the end of treatment. Women of childbearing potential must not rely on hormone-containing contraceptives as a form of birth control during the study. Female subjects using a hormone containing contraceptive prior to screening may continue their contraceptive regimen in addition to the study specified methods of birth control.
   * intrauterine device (IUD) with a documented failure rate of less than 1% per year
   * female barrier method: cervical cap or diaphragm with spermicidal agent
   * tubal sterilization
   * vasectomy in male partner
8. Subjects must be of generally good health as determined by the investigator.
9. Subjects must be able to comply with the dosing instructions for study drug administration and be willing to complete the study schedule of assessments.

Exclusion Criteria:

1. Pregnant or nursing female
2. Current or prior history of clinical hepatic decompensation (e.g., ascites, encephalopathy or variceal hemorrhage, model for end-stage liver disease (MELD)<12)
3. Prior treatment for hepatitis C virus infection
4. Infection with hepatitis B virus (HBsAg positive)
5. Chronic use of systematically administered immunosuppressive agents (e.g., prednisone equivalent >10 mg/day)
6. Use of any prohibited concomitant medications within 28 days of the Baseline/Day 1 visit.
7. Contraindications to PEG
8. Known hypersensitivity to the metabolites or formulation excipients of PEG (for Arm 1 subjects)
9. Active significant psychiatric condition(s) including severe depression, severe bipolar disorder and schizophrenia. Other psychiatric disorders are permitted if the condition is well controlled with a stable treatment regimen for ≥ 1 year from screening, or inactive for ≥ 1 year from screening.
10. Presence of autoimmune disorders (e.g., systemic lupus erythematosus, rheumatoid arthritis, sarcoidosis, psoriasis of greater than mild severity)
11. History of clinical significant retinal disease
12. Clinical evidence of cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Mehta, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- YR Gaitonde Centre for AIDS Education and Johns Hopkins University Collaborative Integrated Care Center (YRG-JHU ICC), Bilāspur, Chhattisgarh, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOF+DAC+PEG | SOF+DAC, DOT | SOF+DAC, Standard
Started | 50 | 50 | 50
Completed | 47 | 45 | 45
Not Completed | 3 | 5 | 5
Not completed — Death | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Incarcerated | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOF+DAC+PEG | SOF+DAC, DOT | SOF+DAC, Standard | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [21 to 31] | 26 [22 to 31] | 25 [21 to 30] | 25 [22 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 50 | 50 | 50 | 150
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indian | 50 | 50 | 50 | 150
Region of Enrollment [Number; unit: participants]
  India | 50 | 50 | 50 | 150
Educational attainment [Count of Participants; unit: Participants]
  None | 3 | 2 | 6 | 11
  Primary school | 19 | 16 | 15 | 50
  Secondary school | 9 | 20 | 17 | 46
  At least high school | 19 | 12 | 12 | 43
Employment [Count of Participants; unit: Participants]
  Monthly wages | 19 | 16 | 12 | 47
  Weekly wages | 5 | 8 | 3 | 16
  Daily wages | 22 | 25 | 28 | 75
  Unemployment | 3 | 1 | 7 | 11
  Missing | 1 | 0 | 0 | 1
Marital status [Count of Participants; unit: Participants]
  Never married | 31 | 32 | 30 | 93
  Currently married | 15 | 13 | 17 | 45
  Separated | 0 | 1 | 0 | 1
  Living with partner | 4 | 4 | 3 | 11
Injection drug use frequency in prior month [Count of Participants; unit: Participants]
  None | 3 | 5 | 4 | 12
  Once a week to less than twice a week | 24 | 17 | 22 | 63
  Twice a week to six times a week | 15 | 15 | 18 | 48
  Daily | 8 | 13 | 6 | 27
Non-injection drug use in prior month [Count of Participants; unit: Participants] | 42 | 38 | 41 | 121
Alcohol use [Count of Participants; unit: Participants]
  No/mild use | 46 | 47 | 45 | 138
  Harmful/hazardous use | 3 | 2 | 5 | 10
  Alcohol dependence | 1 | 1 | 0 | 2
Depressive symptoms [Count of Participants; unit: Participants]
  None | 37 | 28 | 31 | 96
  Mild | 10 | 17 | 15 | 42
  Moderate | 3 | 5 | 3 | 11
  Moderately severe to severe | 0 | 0 | 1 | 1
Quality of life [Median (Inter-Quartile Range); unit: Self-rated health scale (0-100))] — Quality of life evaluated using the Euro-Quality of life - 5 Dimensions (EQ5D) scale. The EQ-5D-5L is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine' with values from 100 to 0. This outcome reported here is based on the EQ VAS which ranges from 0 to 100
  Self-rated health scale (0-100)) | 90 [80 to 100] | 78 [50 to 95] | 80 [60 to 96] | 80 [60 to 100]
HIV-infected [Count of Participants; unit: Participants] | 0 | 1 | 0 | 1
Median HCV RNA [Median (Inter-Quartile Range); unit: log 10 copies/ml] | 5.4 [4.1 to 6.3] | 5.6 [4.3 to 6.2] | 5.7 [5.1 to 6.5] | 5.6 [4.4 to 6.3]
Median calculated fibrosis score (FIB-4) [Median (Inter-Quartile Range); unit: units on a scale] — Fibrosis-4 (FIB-4) is a non-invasive Marker of Hepatic Fibrosis: Fibrosis-4 (FIB-4). Fibrosis-4 is the ratio of age in years and aminotransferase to platelet count. It is a non-invasive hepatic fibrosis index score combining standard biochemical values, platelets, alanine aminotransferase (ALT), AST and age that is calculated using formula: FIB-4 = (Age [years] x AST [U/L]) / (platelets [10^9/L] x (square root of ALT [U/L])). A FIB-4 index of < 1.45 indicated no or moderate fibrosis and an index of > 3.25 indicated extensive fibrosis/cirrhosis.
  units on a scale | 0.69 [0.51 to 0.88] | 0.68 [0.47 to 1.12] | 0.73 [0.54 to 1.14] | 0.68 [0.49 to 1.08]

OUTCOME MEASURES:

1. Primary Outcome: SVR12
Description: Percentage of participants achieving sustained virologic response 12 weeks quantification) after treatment is completed (SVR12) as assessed by HCV RNA less than the lower limit of quantification measured 12 weeks after treatment completion
Time Frame: 12 weeks after treatment completion, 16 weeks for SOF+DAC+PEG and 24 weeks for SOF+DAC
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+DAC+PEG | SOF+DAC, DOT | SOF+DAC, Standard
Number analyzed (Participants) | 50 | 50 | 50
Participants | 26 | 30 | 17

2. Secondary Outcome: Serious Adverse Events
Description: Number of participants with treatment-related serious adverse events by laboratory tests and physician examination
Time Frame: 16 weeks for SOF+DAC+PEG and 24 weeks for SOF+DAC
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+DAC+PEG | SOF+DAC, DOT | SOF+DAC, Standard
Number analyzed (Participants) | 50 | 50 | 50
Participants | 0 | 0 | 0

3. Secondary Outcome: Medication Adherence
Description: Adherence to medication regimen defined using a combination of the biometric data for Arms 1 and 2 and self-report and pill counts for Arm 3. Percentage reporting at least 90% adherence
Time Frame: 4 weeks for SOF+DAC+PEG and 12 weeks for SOF+DAC
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+DAC+PEG | SOF+DAC, DOT | SOF+DAC, Standard
Number analyzed (Participants) | 50 | 50 | 50
Participants | 35 | 31 | 10

ADVERSE EVENTS:
Time Frame: 16 weeks for Arm 1 and 24 weeks for ARms 2 and 3
Arm/Group | SOF+DAC+PEG | SOF+DAC, DOT | SOF+DAC, Standard
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Adherence measurements differ by arm (Arm 1 and 2 included daily observation of doses). Adherence assessment for Arm 3 based on participant completing a visit to pick up medication refill.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT03480932/Prot_SAP_000.pdf